CLINICAL TRIAL: NCT04685772
Title: Assessment of the Efficacy of Medrol Dose Pack for Post-Concussive Headaches
Brief Title: Assessment of the Efficacy of Medrol Dose Pack for Acute Post-Concussive Headaches
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1092
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Post-Concussion Syndrome; Headache
Keywords: Methylprednisolone; Medrol Dose Pack; Steroid
MeSH Terms: conditions — Post-Concussion Syndrome; Headache | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Methylprednisolone — The Methylprednisolone dose pack (Medrol Dose Pack) is pre-packaged with dosing instructions. This dose pack is tapered over 7 days and administration will be the following for all patients:
  Day 1 (total 24 milligrams (mg)) - 8mg before breakfast, 4mg after lunch and dinner, and 8mg at bedtime Day 2 (total 20mg) - 4mg before breakfast, after lunch and dinner, and 8mg at bedtime Day 3 (total 16mg) - 4mg before breakfast, lunch, dinner, and at bedtime Day 4 (total 12mg) - 4mg before breakfast, after lunch, and at bedtime Day 5 (total 8mg) - 4mg before breakfast and at bedtime Day 6 (total 4mg) - 4mg before breakfast Day 7 (total 0mg) - Completed
  Other Names: No methylprednisolone

SUMMARY:
This novel pilot project will assess the effectiveness of corticosteroids in treatment of acute post-concussion headache. The investigators hypothesize that the use of corticosteroids will cause significant headache reduction in frequency and/or intensity than individuals who undergo the current standard of care. Additionally, the investigators hypothesize that corticosteroid use will lead to a reduction in other somatic symptoms including vestibular symptoms, leading to quicker return to school, work, and/or ability to play sports.

DETAILED DESCRIPTION:
To the best of the investigators' knowledge, this is a novel study. Studies have been previously done on individuals who have suffered an acute TBI and were admitted to an intensive care unit (ICU) setting but none have been completed on individuals who suffer post-concussion headaches. Despite a high prevalence of post-concussive headache, there are no evidence-based guidelines for acute or preventive pharmacological treatment. Patients who experience very frequent or daily headache post-concussive headache are also at risk of developing medication-overuse headache (MOH)12. In addition, patients with post-concussive headache experience disabling comorbidities such as symptoms of depression, anxiety, and sleep disturbances 12 This study will be of benefit to patients who suffer headaches after a concussion because, though various treatments have been studied, including a combination of Reglan and Benadryl (63% effective in one prospective study) triptans vs non-triptans (70% effective vs 42% effective in one retrospective trial), gabapentin vs tricyclic antidepressants vs. no medication (no significant difference in outcome), none have been established as a definitive treatment regimen for post-concussive headache 12. Corticosteroids are currently utilized for management of these headaches; they are done so at the discretion of the physician and like the aforementioned medications, are not standard of care. Corticosteroid used in severe TBI (GCS < 8) have been widely studied8, however the utility has not been conclusive. Of note, case studies in the pediatric population with mild TBI (GCS 13-15) and post-concussive headache, report that they respond well to the Medrol Dose Pack with headache improvement during or after completion of the medication2. Currently, there is no standard treatment of post-concussion headaches, and in clinical practice, it has been observed that only approximately 50% of patients improve without any medication use. It is important to establish the role of corticosteroids in treating post-concussive headaches because they may improve quality of life and accelerate patient's functional recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (in person or via telehealth)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged >18 years old
4. Ability to take oral medication and be willing to adhere to the study regimen as described in this protocol
5. Patients presenting with all types of post-concussive headache with >5/10 in severity on the numerical analog scale.
6. Headache that occurs for > 4 hours per day
7. Headache that occurs every day
8. Headache that began after concussion, patient was diagnosed at an outpatient clinic or was hospitalized
9. Headache developed within 7 days post-injury and patient presenting within 30 days from initial trauma
10. A diagnosis of concussion.
11. If a patient is taking another pain medication, this still be included in the stud

Exclusion Criteria:

1. Any evidence of known intracranial hemorrhage on neuroimaging
2. Headache developing after 7 days post injury and patient presenting after 30 days from initial trauma
3. Headache occurs < 4 hours per day
4. Headache does not occur daily
5. Age < or = 18
6. Headache is < 5 in severity on numerical analog scale
7. Presence of increase in intracranial pressure or papilledema
8. Any contraindication to corticosteroids
9. Allergy or sensitivity to corticosteroids
10. Active Tuberculosis
11. Active pregnancy
12. Currently on corticosteroids for another reason
13. Participants with fungal infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusion criteria will be consented for the study. Patients will be recruited when they follow up on their initial appointment after hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in headaches | 1 Week
  Defined as change in headache in response to medication

SECONDARY OUTCOMES:
Change in total Post Concussion Symptom (0-120) scores over time | 12 weeks
  change in the NEW total PCSS score from baseline (day0) to week 1, to week 4 and to week 12; Higher scores indicate worse symptoms.
EQ-5D (Euro Qual Health State Questionnaire) score changes (1-100 in each category); higher score indicates better state of health in several domains. | 12 weeks
  EQ-5D score in the categories of 'Usual Activities' and 'Pain/Discomfort' of the EQ-5D Health Questionnaire between visit 1 (day 7) and visit 5(week 11/12)
Diary of other medication use and pain level | 12 weeks
  Secondary outcome 9: Each patient will be asked to keep a daily diary, recording pain medications used and a pain level (in a scale of 0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Jamie S Ullman, MD, Principal Investigator — Hofstra Northwell School of Medicine
Locations (1):
- Northwell Health - North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bulamu NB, Kaambwa B, Ratcliffe J. A systematic review of instruments for measuring outcomes in economic evaluation within aged care. Health Qual Life Outcomes. 2015 Nov 9;13:179. doi: 10.1186/s12955-015-0372-8. PMID 26553129
- [Background] Bramley H, Hong J, Zacko C, Royer C, Silvis M. Mild Traumatic Brain Injury and Post-concussion Syndrome: Treatment and Related Sequela for Persistent Symptomatic Disease. Sports Med Arthrosc Rev. 2016 Sep;24(3):123-9. doi: 10.1097/JSA.0000000000000111. PMID 27482778
- [Background] Bramley H, Melinosky C, Silvis M, Ross S. Pediatric posttraumatic headache: two cases using steroids as abortive therapy. Pediatr Emerg Care. 2012 Oct;28(10):1081-4. doi: 10.1097/PEC.0b013e31826ceeeb. PMID 23034499
- [Background] Cushman DM, Borowski L, Hansen C, Hendrick J, Bushman T, Teramoto M. Gabapentin and Tricyclics in the Treatment of Post-Concussive Headache, a Retrospective Cohort Study. Headache. 2019 Mar;59(3):371-382. doi: 10.1111/head.13451. Epub 2018 Nov 19. PMID 30451286
- [Background] Ducic I, Sinkin JC, Crutchfield KE. Interdisciplinary treatment of post-concussion and post-traumatic headaches. Microsurgery. 2015 Nov;35(8):603-7. doi: 10.1002/micr.22503. Epub 2015 Sep 26. PMID 26409037
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Halstead ME. Pharmacologic Therapies for Pediatric Concussions. Sports Health. 2016 Jan-Feb;8(1):50-2. doi: 10.1177/1941738115622158. PMID 26660460
- [Background] Hoshide R, Cheung V, Marshall L, Kasper E, Chen CC. Do corticosteroids play a role in the management of traumatic brain injury? Surg Neurol Int. 2016 Sep 13;7:84. doi: 10.4103/2152-7806.190439. eCollection 2016. PMID 27656315
- [Background] Kacperski J. Pharmacotherapy for Persistent Posttraumatic Headaches in Children and Adolescents: A Brief Review of the Literature. Paediatr Drugs. 2018 Oct;20(5):385-393. doi: 10.1007/s40272-018-0299-8. PMID 29876872
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Background] Kuczynski A, Crawford S, Bodell L, Dewey D, Barlow KM. Characteristics of post-traumatic headaches in children following mild traumatic brain injury and their response to treatment: a prospective cohort. Dev Med Child Neurol. 2013 Jul;55(7):636-41. doi: 10.1111/dmcn.12152. Epub 2013 Apr 5. PMID 23560811
- [Background] Larsen EL, Ashina H, Iljazi A, Al-Khazali HM, Seem K, Ashina M, Ashina S, Schytz HW. Acute and preventive pharmacological treatment of post-traumatic headache: a systematic review. J Headache Pain. 2019 Oct 21;20(1):98. doi: 10.1186/s10194-019-1051-7. PMID 31638888
- [Background] Marshall S, Bayley M, McCullagh S, Velikonja D, Berrigan L, Ouchterlony D, Weegar K; mTBI Expert Consensus Group. Updated clinical practice guidelines for concussion/mild traumatic brain injury and persistent symptoms. Brain Inj. 2015;29(6):688-700. doi: 10.3109/02699052.2015.1004755. Epub 2015 Apr 14. PMID 25871303
- [Background] Potter S, Leigh E, Wade D, Fleminger S. The Rivermead Post Concussion Symptoms Questionnaire: a confirmatory factor analysis. J Neurol. 2006 Dec;253(12):1603-14. doi: 10.1007/s00415-006-0275-z. Epub 2006 Oct 24. PMID 17063314
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Seifert T. Post-Traumatic Headache Therapy in the Athlete. Curr Pain Headache Rep. 2016 Jun;20(6):41. doi: 10.1007/s11916-016-0568-6. PMID 27184059
- [Background] Solomon S. Post-traumatic headache: commentary: an overview. Headache. 2009 Jul;49(7):1112-5. doi: 10.1111/j.1526-4610.2009.01462.x. PMID 19583600
- [Background] Bland JM, Altman DG. Applying the right statistics: analyses of measurement studies. Ultrasound Obstet Gynecol. 2003 Jul;22(1):85-93. doi: 10.1002/uog.122. PMID 12858311
- See also: Medrol Dose Pack Product information — https://reference.medscape.com/drug/medrol-medrol-dosepak-methylprednisolone-342746